CLINICAL TRIAL: NCT05901129
Title: The Efficacy of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) on Postoperative Pain and Total Analgesic Consumption in Patients Undergoing Shoulder Surgery
Brief Title: The Efficacy of SPSIPB on Postoperative Pain in Patients Undergoing Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Assisstant Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SPSIPB on shoulder surgery
Record Dates: First submitted 2023-06-01; First posted 2023-06-13 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Post Operative Pain
Keywords: serratus posterior superior intercostal plane block; postoperative pain; shoulder surgery; regional anesthesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIPB (Active Comparator): SPSIP block is the intervention used in this study. It was performed when the patient is in lateral decubitis position. A high frequency (7-12 MHz) linear transducer of the ultrasound device is placed at the spinae scapula level in the transverse plane, and the upper medial border of the scapula, the trapezius muscle, rhomboid muscle, serratus posterior superior muscle (SPSM) and the second and third ribs are visualized. The sonovisible needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs in order to reach the fascial plane between the SPSM and intercostal muscles. After contact of the needle with the rib gently, and a total of 30 mL of 0.25% bupivacaine is administered to the superficial to the intercostal muscle. All patients had 3x400 mg ibuprofen intravenous (i.v.) in postoperative 24 hours. 50 mg tramadol was given as a rescue analgesic drug to the patients who had numerical rating scale (NRS) 4 or higher.
  Interventions: Other: Serratus posterior superior intercostal plane block (SPSIPB)
- Control (No Intervention): Control group patients were not subjected to any block or local infiltration anesthesia (local anesthetic administration around the incision). Their postoperative pain was relieved with ibuprofen 3x400mg intravenous (i.v.) in postoperative 24 hours. The patients had NRS score 4 or higher were given 50 mg tramadol as a rescue analgesic.

INTERVENTIONS:
Other: Serratus posterior superior intercostal plane block (SPSIPB) — Serratus posterior superior intercostal plane block is the intervention used in this study. It was performed when the patient is in lateral decubitis position. A high frequency (7-12 MHz) linear transducer of the ultrasound device is placed at the spinae scapula level in the transverse plane, and the upper medial border of the scapula, the trapezius muscle, rhomboid muscle, serratus posterior superior muscle (SPSM) and the second and third ribs are visualized. The sonovisible needle is then advanced immediately medial to the scapula, aiming for the area between the second and third ribs in order to reach the fascial plane between the SPSM and intercostal muscles. After contact of the needle with the rib gently, 1-2mL of saline is used to confirm the correct plane, and a total of 30 mL of 0.25% bupivacaine is administered to the superficial to the intercostal muscle.
  Arms: SPSIPB

SUMMARY:
Aim is to assess the postoperative analgesic efficacy of SPSIPB and its effect on opioid consumption in patients undergoing shoulder surgery.

DETAILED DESCRIPTION:
There were three randomized groups: Group 1 (no block-control group, n=12) Group 2 (SPSIPB-2nd rib targetted, n=12), Group 3 (SPSIPB-3rd rib targetted, n=12). All patients had standard general anesthesia. Group 2 and Group 3 had serratus posterior superior intercostal plane block (SPSIPB) with 0.25% bupivacaine (total volume of 30 ml) before the surgery. Local anesthetic was injected between 2nd rib an serratus posterior superior muscle in Group 2 and it was injected between 3rd rib and same muscle in Group 3. All patients had 50 mg dexketoprofen and 1 gr paracetamol intravenos (i.v.) 10 minutes prior to skin closure. All patients had ibuprofen 3x400 mg in postoperative 24 hours. Numerical rating scale (NRS) was used to assess postoperative pain on 1st, 6th, 12th, 18th and 24th hour after the surgery. 50 mg tramadol was administered as a rescue analgesic in all patients.Total tramadol consumption was calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent open or arthroscopic shoulder surgery under general anesthesia and were American Society of Anesthesiologists (ASA) I-II-III according to the ASA risk classification.

Exclusion Criteria:

* Patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Total tramadol consumption | Postoperative 24 hours
  Postoperative total analgesic need was recorded as "milligram" in unit.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093